CLINICAL TRIAL: NCT06531616
Title: Healthcare Professionals' Attitudes, Knowledge, and Behaviours Toward Clinical Research in the United Arab Emirates
Brief Title: Healthcare Professionals' Attitude Towards Clinical Research in the United Arab Emirates
Status: Completed | Type: Observational
Sponsor: Abu Dhabi Health Services Company (Other Government)
Responsible Party: Principal Investigator, Alina Naeem, Assistant Manager Research Performance, Abu Dhabi Health Services Company
Other Study IDs: AbuDhabiHealthSvsCo
Record Dates: First submitted 2024-07-26; First posted 2024-08-01 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Behavior, Consumer; Research, Communication; Knowledge, Attitudes, Practice
Keywords: Healthcare Professionals; Allied Health; Doctor; Nurses; Clinical Research
MeSH Terms: conditions — Consumer Behavior; Communication; Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare professionals working at SEHA: SEHA Healthcare employees (doctors, nurses, and allied health staff) will be approached through email to answer the study survey.

SUMMARY:
Abu Dhabi Health Services Company (SEHA) is already in the process of providing support for research infrastructure, such as trained staff, medical facilities, funding, and training needs for its healthcare professionals (HCPs). An HCP's own interest in clinical research is an individualistic trait that SEHA wants to target and develop, complementary to its medical staff specialty, educational background, and willingness to learn.

The investigators' aim with this study is to understand the participants' perspective on challenges and barriers stopping them from conducting research and what supportive measures they have around them from the organization and the United Arab Emirates (UAE) that back their growth as research professionals at SEHA.

DETAILED DESCRIPTION:
The investigators' aim with this study is to understand healthcare professionals' (HCPs) perspective on challenges and barriers stopping them from conducting research and what supportive measures they have around them from the organization and the United Arab Emirates (UAE) that back their growth as research professionals at Abu Dhabi Health Services Company -SEHA.

Investigators hypothesize that participants will give positive feedback on their interest in conducting clinical research but will outline barriers like lack of training opportunities, trained clinical operations staff, organizational support, protected time, etc. Moreover, they will also highlight the lack of data system training, participant accrual challenges, software interoperability issues, sponsor and contract research organization (CRO) issues, and lack of funding opportunities as major barriers to conducting research in the UAE.

ELIGIBILITY:
Inclusion Criteria:

* Current SEHA Employee
* Identify as a Healthcare Professional

Exclusion Criteria:

* Non-SEHA individuals
* Non-Healthcare professionals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of SEHA healthcare employees.
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Understanding Knowledge and Attitudes of SEHA Healthcare professionals toward clinical research. | 3 months
  A self-built survey was created to cover the different aspects of the United Arab Emirates (UAE) healthcare organizational practices and clinical research practices. The survey was pilot-tested on 6 volunteers not related to the Abu Dhabi Health Services Company (SEHA) for comprehension and ease of reading. The survey aims to understand participants' perspectives on challenges and barriers stopping them from conducting research and what supportive measures they have around them from the SEHA as an organization and the UAE that back their growth as medical research professionals. The data collected can help guide in bringing positive organizational changes to enhance clinical research at SEHA and in the UAE.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam S Al Harbi, MD, Study Chair — Abu Dhabi Health Services Co. -SEHA; Erik BS Koornneef, PHD, Study Chair — Abu Dhabi Health Services Co. -SEHA
Locations (1):
- SEHA Head Quaters-Reserach Department, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Hajri A, Al-Khabori M, Rasool W. Productivity of Clinical Trials Conducted in the Gulf Cooperative Council Region. Sultan Qaboos Univ Med J. 2022 Nov;22(4):501-507. doi: 10.18295/squmj.11.2021.144. Epub 2022 Nov 7. PMID 36407711
- [Result] D'Arrietta LM, Vangaveti VN, Crowe MJ, Malau-Aduli BS. Rethinking Health Professionals' Motivation to Do Research: A Systematic Review. J Multidiscip Healthc. 2022 Jan 26;15:185-216. doi: 10.2147/JMDH.S337172. eCollection 2022. PMID 35115782
- [Result] Ito-Ihara T, Hong JH, Kim OJ, Sumi E, Kim SY, Tanaka S, Narita K, Hatta T, Choi EK, Choi KJ, Miyagawa T, Minami M, Murayama T, Yokode M. An international survey of physicians regarding clinical trials: a comparison between Kyoto University Hospital and Seoul National University Hospital. BMC Med Res Methodol. 2013 Oct 25;13:130. doi: 10.1186/1471-2288-13-130. PMID 24156760
- [Result] Silberman EK, Belitsky R, Bernstein CA, Cabaniss DL, Crisp-Han H, Dickstein LJ, Kaplan AS, Hilty DM, Nadelson CC, Scheiber SC. Recruiting researchers in psychiatry: the influence of residency vs. early motivation. Acad Psychiatry. 2012 Mar 1;36(2):85-90. doi: 10.1176/appi.ap.10010010. PMID 22532195
- See also: Comparison of the Perceptions between Investigators and Clinical Research Associates in Role Performances of Clinical Research Coordinators — https://doi.org/10.5762/KAIS.2014.15.8.5095
- See also: The Challenges In Conducting Research Studies In Arabic Countries — http://dx.doi.org/10.2147/OAJCT.S215738